CLINICAL TRIAL: NCT00005628
Title: A Phase II Trial of Active Specific Immunotherapy in Patients With Recurrent Soft Tissue Sarcoma Using Autologous Tumor-derived Heat Shock Protein-Peptide Complex (HSPPC-96)
Brief Title: Vaccine Therapy in Treating Patients With Recurrent Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 99-077; CDR0000067781 (Registry Identifier: PDQ (Physician Data Query)); NCI-H00-0052
Record Dates: First submitted 2000-05-02; First posted 2004-04-02 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Sarcoma
Keywords: recurrent adult soft tissue sarcoma; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma | interventions — vitespin

INTERVENTIONS:
Biological: vitespen

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells.

PURPOSE: Phase II trial to study the effectiveness of vaccine therapy in treating patients who have recurrent soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of autologous tumor cell-derived heat shock protein peptide vaccine in terms of the rate of complete and partial response and time to progression in patients with recurrent soft tissue sarcoma. II. Determine the safety and tolerability of this treatment regimen in this patient population. III. Determine the anti-tumor response to this treatment regimen in these patients.

OUTLINE: At approximately 5 weeks after surgery, patients receive autologous tumor cell-derived heat shock protein peptide vaccine intradermally weekly for 4 weeks. Patients receive subsequent vaccinations once every 2 weeks for at least 12 weeks in the absence of disease progression or unacceptable toxicity. Patients with improving or stable disease or without recurrence continue on therapy for up to 1 year.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed recurrent soft tissue sarcoma Incompletely or completely resected metastatic or locally recurrent disease (surgery must be performed with intent of complete resection) No active brain metastases

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: Karnofsky 70-100% Life expectancy: At least 16 weeks Hematopoietic: WBC at least 3,000/mm3 Absolute neutrophil count at least 1,000/mm3 Platelet count at least 80,000/mm3 Hepatic: Not specified Renal: Creatinine no greater than 2.5 mg/dL Cardiovascular: No New York Heart Association class III or IV heart disease Other: No active infections requiring antibiotics within 2 weeks of study No other serious medical illness requiring hospitalization No history of primary or secondary immunodeficiency or autoimmune disease No contraindications to MRI (e.g., aneurysm clips or cardiac pacemakers) Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 6 weeks since prior immunotherapy and recovered Chemotherapy: At least 6 weeks since prior chemotherapy and recovered Endocrine therapy: No concurrent systemic corticosteroids Radiotherapy: At least 6 weeks since prior radiotherapy and recovered Surgery: See Disease Characteristics No prior splenectomy Other: At least 6 weeks since other prior experimental anticancer therapy and recovered No concurrent non-steroidal anti-inflammatory drugs or other immunosuppressive drugs No other concurrent participation in a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-11; Primary Completion 2001-08 (Actual); Study Completion 2001-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Maki, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States